CLINICAL TRIAL: NCT00734981
Title: Efficacy Evaluation of a Novel Diagnostic Assay Which is the Basis for Seaforia Diagnostic System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lotus Bio Inc. (Other)
Responsible Party: Kahana Arik MD., Assuta Medical Centers Ltd.
Other Study IDs: LBI-02-V2
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Male Fertility

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: None Retained — Semen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Evaluation of specificity and sensitivity of Seaforia- an vitro diagnostic system for evaluating semen quality.

DETAILED DESCRIPTION:
Quantities assessment of semen quality as defined by:

Semen volume, semen pH, leukocytes concentration, sperm cells concentration, motile sperm cell concentration, total motile sperm cells threshold and sperm cells morphology

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* 20<Age<45
* Male

Exclusion Criteria:

None

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Semen Quality as determined by the following parameters: Semen volume | The same day as sevan evaluation according to the gold standard
Semen pH | The same day as sevan evaluation according to the gold standard
Leukocytes concentration | The same day as sevan evaluation according to the gold standard
Sperm cells concentration | The same day as sevan evaluation according to the gold standard
Motile sperm cell concentration | The same day as sevan evaluation according to the gold standard
Total motile sperm cells threshold | The same day as sevan evaluation according to the gold standard
Sperm cells morphology | The same day as sevan evaluation according to the gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Centers Ltd., Tel Aviv, Israel